CLINICAL TRIAL: NCT02080975
Title: Determination of Catheter Contact by Evaluation of Microelectrode Near-Field Signals
Acronym: IN-CONTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David B. De Lurgio (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, David B. De Lurgio, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00071344
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Catheter Ablation; Atrial Flutter; Cardiac Arrhythmias
MeSH Terms: conditions — Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Data Collection During Atrial Flutter Ablation (Experimental)
  Interventions: Other: Data Collection During Atrial Flutter Ablation

INTERVENTIONS:
Other: Data Collection During Atrial Flutter Ablation — All enrolled patients are clinically indicated for an atrial flutter ablation. The patients who consent for this study will have additional electrocardiograms taken during their procedure for future review, as well as ultrasound images form inside their heart. This will lengthen the ablation by approximately 10 minutes, but is not a separate procedure.

SUMMARY:
Successful radio frequency (RF) cardiac catheter ablation requires the creation of lesions by delivering energy while maintaining adequate catheter contact with the endocardium. Unfortunately, it is difficult to identify contact intraoperatively as a typical RF ablation catheter lacks clear indications of contact. We propose to use the Boston Scientific IntellaTip MiFi catheter to explore whether characteristics of the electrograms produced by the mini-electrodes on the ablation tip could help confirm tissue contact. Using an ultrasound catheter to define instances of clear contact and non-contact, we will determine whether the micro-electrodes produce sufficient information to confirm catheter contact. We propose that the MiFi catheter produces sufficient signal characteristics that can be used as an effective surrogate for adequate tissue contact.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of typical atrial flutter
* Subject is clinically indicated for right sided atrial flutter ablation
* Patient is willing and able to understand and sign the informed consent document
* Patient is over 18 years of age
* Patient is willing and able to comply with the study protocol

Exclusion Criteria:

* Patient has one of the following cardiac comorbidities: hypertrophic cardiomyopathy, structural heart disease, congestive heart failure
* Patient has history of the following arrhythmias: ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White syndrome
* Patient has a contraindication to right atrium ablation, including but not limited to: right atrial thrombus, active systemic infection, or a coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation between catheter contact and micro electrode signals | During Procedure
  The known contact state of the ablation catheter will be compared in a blinded fashion to the signals from the microelectrodes to determine if a relationship exits.

SECONDARY OUTCOMES:
Document the electrogram signatures that help demonstrate catheter tip contact | During Procedure

CONTACTS AND LOCATIONS:
Overall Officials: David B De Lurgio, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No